CLINICAL TRIAL: NCT03450915
Title: A Pivotal Multi-center, Randomized, Modified Double-blind, Placebo-controlled Phase 3 Trial to Assess the Safety and Clinical Efficacy of M-001 Influenza Vaccine Administered Intra-muscularly Twice in Older Adults and Elderly (≥50 Years).
Brief Title: A Pivotal Trial to Assess the Safety and Clinical Efficacy of the M-001 as a Standalone Universal Flu Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BiondVax Pharmaceuticals ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BVX-010
Record Dates: First submitted 2018-02-08; First posted 2018-03-01 (Actual); Results first posted 2021-09-13 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Influenza
Keywords: Influenza; vaccine; universal; M-001; Multimeric-001; Flu
MeSH Terms: conditions — Influenza, Human | interventions — PN M001; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Experimental group: 2 immunizations with M-001 Control group: 2 injection of saline (placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties are blinded except for the person who prepares the syringe for injection. The M-001 is cloudy white and its appearance is different from the transparent saline that is used for placebo. The person prepares the syringe with an opaque sticker that fully covers the syringe contents. People administering the syringe are not involved or present during syringe preparation, and are thus fully blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-001 (Experimental): Participants will be vaccinated with 1mg dose of M-001 twice: Once at Day 0, and once at Day 21.
  Interventions: Biological: M-001
- Saline (Placebo Comparator): Participants will be vaccinated with saline twice: Once at Day 0, and once at Day 21.
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: M-001 — A recombinant protein containing 9 conserved epitopes from Influenza A and B that are common to the vast majority of influenza viruses.
  Other Names: Multimeric-001
  Arms: M-001
Biological: Saline — 0.9% sodium chloride (NaCl)
  Arms: Saline

SUMMARY:
The pivotal Phase 3 trial plans to enroll a total of approximately 12,460 participants aged 50+ over two years. Participants will be immunized twice with the M-001 universal influenza vaccine candidate or placebo and then followed for up to 2 seasons. The trial will evaluate the number of influenza cases in each group and the severity of illness during the follow up period.

DETAILED DESCRIPTION:
The placebo-controlled pivotal clinical efficacy Phase 3 trial plans to enroll a total of approximately 12,460 participants over two years. Participants will be immunized twice with the M-001 influenza vaccine candidate or placebo. Influenza incidence and illness severity will be evaluated throughout the follow-up period of up to two years. Participants will be 50 years and older, with at least half over 65 years of age.

The trial is expected to take place in eastern European countries and begin prior to the 2018/19 Northern Hemisphere flu season.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 50 years of age (inclusive) or older, mentally competent, willing and able to give the written informed consent prior to study entry
2. Able to comply with the trial procedures and be available for all study visits.
3. Medically stable. (Subjects may have underlying chronic conditions such as hypertension, diabetes, ischemic heart disease, or hypothyroidism, as long as their symptoms/signs are controlled. If they are on medication for a condition, the medication dose must have been stable for at least 3 months preceding vaccination).
4. Women of childbearing potential (not surgically sterile or postmenopausal for greater than or equal to one year) and men must agree to practice adequate contraception (barrier or hormone methods or intra uterine device (IUD) for women and a condom for men) throughout the study treatment and for at least up to day 51 (for female) and day 111 (for male) of the trial (i.e. 30 (for female) and 90 (for male) days after the last dose of the IMP)
5. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study vaccination.

Exclusion Criteria:

1. History of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine.
2. Known or suspected (or have a high risk of developing) impairment/alteration of immune function (excluding that normally associated with advanced age).
3. Receipt of: a) Immunosuppressive drugs: i) systemic glucocorticoids >/= 10 mg prednisone per day ii) cytotoxic drugs b) Investigational drugs within 30 days before, or planned during, the study c) Blood products within 3 months before, or planned during, the study d) Influenza vaccine within 6 months before the study) Other vaccines within 30 days before, or planned during, the study
4. Any serious disease such as: cancer, autoimmune disease, advanced arteriosclerotic disease or complicated diabetes mellitus, chronic obstructive pulmonary disease (COPD) that requires oxygen therapy, acute or progressive hepatic disease, acute or progressive renal disease, or congestive heart failure, as judged by the PI.
5. An acute illness, including an axillary temperature greater than 38 Celsius (38ºC), occurred within 1 week before first vaccination
6. Positive positive urine pregnancy test prior to vaccination or women who are breastfeeding.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12460 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Ben-Yedidia, PhD, Study Director — BiondVax Pharmaceuticals ltd.
Locations (2):
- Poland (2):
  - Jagiellońskie Centrum Innowacji Sp.z o.o., Krakow, Ul. Bobrzyńskiego 14,
  - Jagiellońskie Centrum Innowacji Sp.z o.o., Krakow

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | M-001 | Saline
Started | 6230 | 6230
Completed | 5827 | 5855
Not Completed | 403 | 375

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is the Intention-to-treat population, i.e. subjects who received at least one vaccination
Groups:
- Total: Total of all reporting groups
Arm/Group | M-001 | Saline | Total
Number analyzed (Participants) | 6229 | 6229 | 12458
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3082 | 3081 | 6163
  >=65 years | 3147 | 3148 | 6295
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (8.7) | 64.6 (8.7) | 64.6 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3454 | 3486 | 6940
  Male | 2775 | 2743 | 5518
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 1 | 3
  White | 6227 | 6228 | 12455
Region of Enrollment [Number; unit: participants]
  Bulgaria | 1751 | 1749 | 3500
  Croatia | 78 | 82 | 160
  Georgia | 258 | 256 | 514
  Hungary | 187 | 184 | 371
  Latvia | 268 | 273 | 541
  Poland | 2740 | 2736 | 5476
  Ukraine | 947 | 949 | 1896

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With qRT-PCR or Culture-confirmed Influenza-like Illness
Description: Prevention of influenza disease by comparing the occurrence of either qRT-PCR or culture confirmed influenza in the M-001 experimental group vs. placebo caused by any influenza A or B virus in association with a protocol defined Influenza Like Illness.
Time Frame: From Day 14 post-second vaccination day to end of influenza season, an average of 4 months per participant per year
Population: Per protocol population comprises all subjects who received both doses of vaccine or placebo and had at least one contact with study staff after 15 days or more upon second vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | M-001 | Saline
Number analyzed (Participants) | 5864 | 5905
Participants
  Both seasons | 160 | 138
  Season 2018/2019: number analyzed (Participants) | 1906 | 1917
  Season 2018/2019 | 74 | 60
  Season 2019/2020: number analyzed (Participants) | 3958 | 3988
  Season 2019/2020 | 86 | 78

2. Primary Outcome: Number of Participants With One or More Serious Adverse Events, New Onset Chronic Illness, and Non-solicited Adverse Events
Description: Number of participants with one or more Serious Adverse Events, New Onset Chronic illness, and Non-solicited Adverse Events assessed during one flu season per participant
Time Frame: From Day 0 to end of study completion by participant which coincides with end of flu season in the respective year, an average of 4 months per participant per year
Population: Safety population comprises all subjects enrolled
Measure: Number; unit: participants
Arm/Group | M-001 | Saline
Number analyzed (Participants) | 6230 | 6230
participants
  Serious Adverse Events | 185 | 177
  New Onset Chronic Illness | 167 | 166
  Non-solicited Adverse Events | 781 | 760

3. Secondary Outcome: Number of Participants With Culture-confirmed Influenza Incidence
Description: Occurrence of culture confirmed influenza in the M-001 experimental group vs. placebo caused by any influenza A or B virus in association with a protocol defined Influenza Like Illness.
Time Frame: From Day 14 post-second vaccination day to end of influenza season, an average of 4 months per participant per year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | M-001 | Saline
Number analyzed (Participants) | 5864 | 5905
Participants | 111 | 96

4. Secondary Outcome: Number of Participants With Reduction of Severity of qRT-PCR or Culture-confirmed Influenza
Description: Assessed by reduction of severity of either qRT-PCR or culture-confirmed influenza illness by the reduction due to M-001 in the average number of days with respiratory or systemic symptoms during the first laboratory-confirmed influenza illness episode.
Time Frame: From Day 14 post-second vaccination day to end of influenza season, an average of 4 months per participant per year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | M-001 | Saline
Number analyzed (Participants) | 5864 | 5905
Participants
  < 7 days | 13 | 12
  >= 7 - 14 days | 94 | 71
  >=14 - 21 days | 29 | 29
  >= 21 days | 24 | 26

5. Secondary Outcome: Number of Participants With Influenza-like Illness Symptoms
Description: Assessment of number of participants having ILI symptoms in the experimental or control group
Time Frame: From Day 14 post-second vaccination day to end of influenza season, an average of 4 months per participant per year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | M-001 | Saline
Number analyzed (Participants) | 5864 | 5905
Participants | 1231 | 1266

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | M-001 | Saline
All-Cause Mortality (participants affected / at risk) | 26/6230 | 29/6230
Serious Adverse Events (participants affected / at risk) | 185/6230 | 177/6230
Other Adverse Events (participants affected / at risk) | 781/6230 | 760/6230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M-001 (N=6230) | Saline (N=6230)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 2 (2) | 0 (0)
Cerebrospinal Fluid Circulation Disorder (Nervous system disorders) | 2 (2) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 2 (2) | 5 (5)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 2 (2) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 3 (3)
Cerebrovascular Insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic Stroke (Nervous system disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ulnar Tunnel Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral Ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage Intracranial (Nervous system disorders) | 0 (0) | 2 (2)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar Insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Reactive Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Calculus Urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis Noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Endometrial Hypertrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Reproductive Tract Disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 27 (29) | 28 (30)
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 9 (10)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 6 (6)
Hypertensive Crisis (Vascular disorders) | 4 (4) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Steal Syndrome (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Bleeding Varicose Vein (Vascular disorders) | 0 (0) | 1 (1)
Circulatory Collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Vascular Occlusion (Vascular disorders) | 0 (0) | 1 (1)
Venous Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myocardial Infarction 6 ( (Cardiac disorders) | 6 (6) | 6 (6)
Cardiac Arrest (Cardiac disorders) | 5 (5) | 2 (2)
Cardiac Failure (Cardiac disorders) | 5 (5) | 2 (4)
Angina Pectoris (Cardiac disorders) | 3 (4) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 3 (3) | 3 (3)
Acute Coronary Syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Angina Unstable (Cardiac disorders) | 2 (2) | 4 (4)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac Failure Chronic (Cardiac disorders) | 2 (2) | 5 (5)
Cardiac Failure Congestive (Cardiac disorders) | 2 (2) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Valve Disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular Insufficiency (Cardiac disorders) | 1 (1) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular Disorder (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 4 (4)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
V (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Thyroiditis Subacute (Endocrine disorders) | 1 (1) | 0 (0)
Posterior Capsule Rupture (Eye disorders) | 0 (0) | 1 (1)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal Mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse Event (General disorders) | 3 (3) | 2 (2)
Death (General disorders) | 2 (2) | 2 (2)
Sudden Death (General disorders) | 1 (1) | 3 (3)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Facial Pain (General disorders) | 0 (0) | 1 (1)
General Physical Health Deterioration (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Sudden Cardiac Death (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 1 (1)
Bile Duct Obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis Chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary Dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis Acute 0 0 (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 16 (16) | 13 (13)
Respiratory Tract Infection (Infections and infestations) | 3 (3) | 0 (0)
Atypical Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia Bacterial (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Bacterial Infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 4 (4)
conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Corona Virus Infection (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis Chronic (Infections and infestations) | 1 (1) | 1 (1)
Abdominal Abscess (Infections and infestations) | 0 (0) | 1 (2)
Anal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Bacterial Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured Coccyx (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectosigmoid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue Neoplasm Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast Cancer Stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dysplastic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M-001 (N=6230) | Saline (N=6230)
Cardiac Failure (Cardiac disorders) | 6 (6) | 5 (7)
Myocardial Infarction (Cardiac disorders) | 6 (6) | 6 (6)
Cardiac Failure Chronic (Cardiac disorders) | 4 (4) | 6 (6)
Myocardial Ischaemia (Cardiac disorders) | 3 (3) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 13 (13) | 13 (13)
Nausea (Gastrointestinal disorders) | 8 (9) | 7 (7)
Abdominal Pain Upper (Gastrointestinal disorders) | 7 (8) | 9 (10)
Abdominal Pain (Gastrointestinal disorders) | 5 (5) | 10 (10)
Abdominal Discomfort (Gastrointestinal disorders) | 2 (2) | 6 (6)
Malaise (General disorders) | 38 (40) | 33 (37)
Pyrexia (General disorders) | 33 (35) | 19 (20)
Chills (General disorders) | 26 (28) | 20 (24)
Injection Site Pain (General disorders) | 21 (22) | 3 (3)
Fatigue (General disorders) | 17 (18) | 15 (16)
Injection Site Bruising (General disorders) | 15 (15) | 13 (13)
Injection Site Erythema (General disorders) | 8 (8) | 2 (2)
Asthenia (General disorders) | 7 (7) | 9 (9)
Nasopharyngitis (Infections and infestations) | 25 (25) | 23 (24)
Pneumonia (Infections and infestations) | 19 (19) | 16 (16)
Rhinitis (Infections and infestations) | 16 (16) | 14 (14)
Upper Respiratory Tract Infection (Infections and infestations) | 16 (16) | 18 (18)
Bronchitis (Infections and infestations) | 13 (13) | 16 (16)
Respiratory Tract Infection (Infections and infestations) | 13 (13) | 8 (9)
Urinary Tract Infection (Infections and infestations) | 12 (12) | 6 (6)
Viral Infection (Infections and infestations) | 9 (10) | 7 (7)
Herpes Zoster (Infections and infestations) | 7 (7) | 1 (1)
Conjunctivitis (Infections and infestations) | 6 (6) | 4 (4)
Blood Pressure Decreased (Investigations) | 12 (14) | 6 (6)
Blood Pressure Increased (Investigations) | 6 (6) | 11 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 77 (84) | 54 (60)
Myalgia (Musculoskeletal and connective tissue disorders) | 28 (30) | 26 (28)
Back Pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 11 (11)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6)
Headache (Nervous system disorders) | 106 (113) | 90 (99)
Dizziness (Nervous system disorders) | 16 (17) | 19 (21)
Irritability (Psychiatric disorders) | 15 (15) | 17 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 57 (60) | 60 (65)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 42 (50) | 55 (57)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 40 (43) | 41 (43)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 33 (35) | 39 (42)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 24 (25) | 20 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 11 (11)
Asthma (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 13 (14)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 26 (28) | 23 (26)
Pruritus (Skin and subcutaneous tissue disorders) | 21 (21) | 17 (17)
Erythema (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 15 (15)
Hypertension (Vascular disorders) | 26 (26) | 29 (30)
Hypertensive Crises (Vascular disorders) | 8 (8) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT03450915/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT03450915/SAP_001.pdf